CLINICAL TRIAL: NCT04226365
Title: Treatment for Post-concussive Headache: A Randomized, Placebo-controlled, Double Blinded Trial
Brief Title: Pediatric Concussion Outcomes
Acronym: PeCon
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped prematurely due to a low enrollment rate.
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-83
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Concussion Post Syndrome; Headaches Posttraumatic; Mild Traumatic Brain Injury
Keywords: concussion; headache; mild TBI; post concussion
MeSH Terms: conditions — Post-Concussion Syndrome; Post-Traumatic Headache; Brain Concussion; Headache | interventions — Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): 10mg capsule once daily for 4 weeks of nortriptyline
  Interventions: Drug: Nortriptyline
- Control (Placebo Comparator): 10mg capsule once daily for 4 weeks of Thick-It filler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nortriptyline — 10mg capsule Nortryptyline
  Other Names: Pamelor
  Arms: Experimental
Drug: Placebo — 10mg capsule Thick-It filler
  Arms: Control

SUMMARY:
This is a randomized, placebo-controlled, double-blinded trial in which subjects with a post concussive headache meeting inclusion criterion will be assigned to one of two treatment groups: placebo or nortriptyline. Each group will be evaluated at week 0 and again each week for the next 4 weeks of treatment with a concussion survey that rates their symptoms. At the end of 4 weeks the study will be unblinded. It is hypothesized that the addition of nortriptyline to the standard headache treatments will result in more rapid decrease of symptom score than with placebo.

DETAILED DESCRIPTION:
Participants are randomly assigned to one of two treatment groups. The experimental group receives standard headache treatment including Tylenol, NSAIDs 2-3x/week, vestibular PT and daily nortriptyline 10mg oral. The control group also receives the standard headache treatment, but will instead be given a placebo, which will look physically identical to the nortriptyline capsule and be comprised of non-active pharmaceutical grade excipient.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Participants aged 13-21 years old
4. In good general health as evidenced by medical history and diagnosed with recent head trauma meeting ICHD-3 criteria for acute posttraumatic headache with symptom onset < 7 days from trauma
5. Ability to take oral medication and be willing to adhere to the medication regimen
6. No loss of consciousness OR loss of consciousness <30 minutes
7. Headache symptoms persisting ≥4 weeks post trauma
8. PCSHE score for headache + pressure in head + neck pain must be > 3
9. After week 4 post-concussion at time of enrollment
10. Not currently receiving pharmacologic treatment for concussion asid from NSAIDs and acetaminophen

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Focal neurological deficits following injury
2. Any acute abnormality on Computed Tomography (if obtained)
3. History of known seizure disorder or moderate or severe TBI
4. Current uncontrolled psychiatric illness given the potential side effects of the study drug (at investigator discretion).
5. Current suicidal ideation as screened for on PHQ on intake
6. A personal history of Brugada syndrome
7. Known allergic reaction to nortriptyline
8. Current pregnancy
9. Positive COVID-19 test in prior 14 days

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Moreno, MD, Principal Investigator — Lancaster General Health Sports Medicine; Laura DiPaolo, MD, Principal Investigator — Lancaster General Health Sports Medicine
Locations (1):
- Penn Medicine Lancaster General Health, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choe MC, Blume HK. Pediatric Posttraumatic Headache: A Review. J Child Neurol. 2016 Jan;31(1):76-85. doi: 10.1177/0883073814568152. Epub 2015 Feb 10. PMID 25670632
- [Background] Kacperski J, Hung R, Blume HK. Pediatric Posttraumatic Headache. Semin Pediatr Neurol. 2016 Feb;23(1):27-34. doi: 10.1016/j.spen.2015.08.005. Epub 2015 Aug 19. PMID 27017019
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] Makdissi M, Schneider KJ, Feddermann-Demont N, Guskiewicz KM, Hinds S, Leddy JJ, McCrea M, Turner M, Johnston KM. Approach to investigation and treatment of persistent symptoms following sport-related concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):958-968. doi: 10.1136/bjsports-2016-097470. Epub 2017 May 8. PMID 28483928
- [Background] Bernard CO, Ponsford JL, McKinlay A, McKenzie D, Krieser D. Do Concussive Symptoms Really Resolve in Young Children? J Head Trauma Rehabil. 2017 Nov/Dec;32(6):413-424. doi: 10.1097/HTR.0000000000000298. PMID 28422893
- [Background] Kuczynski A, Crawford S, Bodell L, Dewey D, Barlow KM. Characteristics of post-traumatic headaches in children following mild traumatic brain injury and their response to treatment: a prospective cohort. Dev Med Child Neurol. 2013 Jul;55(7):636-41. doi: 10.1111/dmcn.12152. Epub 2013 Apr 5. PMID 23560811
- [Background] Johnson JG, Harris ES, Spitzer RL, Williams JB. The patient health questionnaire for adolescents: validation of an instrument for the assessment of mental disorders among adolescent primary care patients. J Adolesc Health. 2002 Mar;30(3):196-204. doi: 10.1016/s1054-139x(01)00333-0. PMID 11869927
- See also: Sport concussion assessment tool - 5th edition — https://doi.org/10.1136/bjsports-2017-097506SCAT5
- See also: Pamelor [package insert]. Hazelwood, MO: Mallinckrodt Inc; 2019. — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=e17dc299-f52d-414d-ab6e-e809bd6f8acb

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Control
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (2) | 14.7 (1) | 14.6 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Post-Concussive Symptom Inventory (PSCI) Score
Description: Post-Concussive Symptom Inventory (PSCI) score of 0-1 on the headache symptom, where the score ranges from 0 (absent) to 6 (severe). A score of 0 is optimal, while a score of 6 is not optimal.
Time Frame: 4 weeks
Population: The trial was terminated before the outcome measure data were collected.
Arm/Group | Experimental | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 39 months
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=4) | Control (N=4)
Headache/Migraine (Nervous system disorders) | 1 (3) | 1 (1)
Sever's Apophysitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT04226365/Prot_SAP_002.pdf
  • Informed Consent Form: English Version (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04226365/ICF_003.pdf